CLINICAL TRIAL: NCT00391638
Title: Pilot Study on Efficacy and Tolerance of Peg-interferon Alpha-2a (Pegasys) Added to Tenofovir DF and Emtricitabine (Truvada) in AGHBe Positive HBV-HIV Co-infected Patients. ANRS HB 01 EMVIPEG.
Brief Title: Efficacy and Tolerance of Peg-interferon Alpha 2a Added to Tenofovir and Emtricitabine in AgHBe Positive HBV-HIV Co-infected Patients
Acronym: HB01EMVIPEG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Gilead Sciences (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004137-15; ANRS HB 01 EMVIPEG
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis B; HIV Infections
Keywords: HIV and Hepatitis B coinfection; Peg interferon; tenofovir; emtricitabine; Hepatitis B e Antigens; Treatment Experienced
MeSH Terms: conditions — Hepatitis B; HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIV antiretroviral therapy, TRUVADA , PEGASYS 180μg (Experimental): Week-8 up Week0: HIV antiretroviral therapy Week 0 up Week 48: HIV antiretroviral therapy + TRUVADA + PEGASYS 180μg Week 48 up Week 72: HIV antiretroviral therapy + TRUVADA Week 72 up Week 144: HIV antiretroviral therapy
  Interventions: Drug: TRUVADA (EMTRICITABINE + TENOFOVIR DF); Biological: PEGASYS 180μg (Interféron pégylé alpha -2a)

INTERVENTIONS:
Drug: TRUVADA (EMTRICITABINE + TENOFOVIR DF) — Truvada ® (200 mg tablet of 300 mg of emtricitabine + tenofovir DF) Dosage 1 tablet taken orally once a day
Biological: PEGASYS 180μg (Interféron pégylé alpha -2a) — Pegasys ® injection 180μg Dosage: A subcutaneous injection per week

SUMMARY:
HBe seroconversion is an important goal for anti-HBV treatment, since it is associated with a non progressive liver infection and a better clinical outcome. However, the rate of HBe seroconversion is low in HIV-HBV co-infected patients, mostly treated by tenofovir and emtricitabine. This study will evaluate the efficacy and the safety of a one-year Peg-interferon alpha 2a additional treatment in patients already treated by tenofovir and emtricitabine without reaching HBe seroconversion.

DETAILED DESCRIPTION:
Many HBV-HIV co-infected patients are currently treated with dual activity drugs such as tenofovir and emtricitabine, often in combination. However, despite the potent antiviral activity of these drugs, the rate of HBe seroconversion is quite low, and not always sustained over time. HBe seroconversion is an important goal for anti-HBV treatment, since it is associated with a non progressive liver infection and a better clinical outcome. On the other hand, treatments with antiviral and immuno-modulator activity such as Peg-interferon, are infrequently used in co-infected patients, despite promising data in the field of HBV mono-infection with increased rates and sustained HBe seroconversions. This pilot study will evaluate the efficacy and the safety of a one-year Peg-interferon alpha 2a additional treatment (180 micro-g once a week, by injection), in 55 patients already treated by tenofovir and emtricitabine for at least 6 months, and who did not reached HBe seroconversion

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Karnofsky above 80 per cent
* Stable ARV since 4 months
* CD4 above 200 per mm3
* ARN VIH below 10000 copies per ml
* hepatitis B chronic with : positive antigenaemia HBe and negative antiHBe, positive DNA HBV before or under tenofovir treatment, DNA HBV negative or below 10000 copies per ml at W-8.
* Previous treatment by tenofovir and lamivudine or emtricitabine more than 6 months

Exclusion Criteria:

* HIV 2 infection
* Hepatitis C or D
* Opportunistic infection
* Alcool consummation more than 50g/d
* Cirrhosis
* Pregnancy or plan of pregnancy
* Breastfeeding
* Immunosuppressive or modulating of the immune response treatment
* Other Hepatitis B treatments than tenofovir, lamivudine or emtricitabine since 6 months
* Malabsorption
* Exclusive HIV therapy with Truvada
* Evolutive cancer under chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients with seroconversion HBe (loose of HBe antigen and acquisition of HBe antibody) and HBV DNA below 2.3 log10 copies per ml | at Week 72

SECONDARY OUTCOMES:
proportion of patients with negative HBe antigen. | at Week 72 and Week 144
proportion of patients with HBV DNA under 2.3 log 10 copies per ml. | at Week 72 and Week 144
proportion of seroconversion HBs. | at Week 72 and Week 144
proportion of patients with no more HBs antigen. | at Week 72 and Week 144
proportion of patients with HBV DNA below 2.3 log 10 copies per ml in relation with 3TC resistance or not before tenofovir treatment; increased of ALT before tenofovir treatment;duration of tenofovir treatment before study. | before tenofovir treatment, duration of tenofovir treatment before study
Biological evolution and histological of hepatic activity and fibrosis. | at day 0 and Week 72
Biochemical response (ALT at normal value). | at Week 72 and Week 144
proportion of patients with :seroconversion HBe and HBV DNA below 2.3 log 10 copies per ml | at Week 48
HBV and HIV resistance mutations to tenofovir DF and Emtricitabine. | at Week 72
Immunological and virological evolution of HIV infection. | between Day 0 and Week 144
Safety | between Day 0 and Week 144
Quality of life | Day 0, Week 12, Week 24, Week 48, Week 72
Treatment adherence | Day 0 to Week 144

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Piroth, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Fabrice Carrat, MD, Study Chair — Inserm U 707 Paris France
Locations (2):
- France (2):
  - Service des Maladies Infectieuses CHU, Dijon
  - Service d'Hépato-Gastroentérologie Hopital Hôtel-Dieu, Lyon